CLINICAL TRIAL: NCT01560143
Title: Pharmacokinetics Of Tigecycline In Morbidly Obese Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Manjunath Prakash Pai (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Manjunath Prakash Pai, Associate Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 11-007; WS2001231 (Other Grant/Funding Number: Pfizer, Inc.)
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tigecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tigecycline (Other): All subjects receive a single dose of tigecycline
  Interventions: Drug: Tigecycline

INTERVENTIONS:
Drug: Tigecycline — 100 mg IV as a single infusion over 30 minutes
  Other Names: Tygacil

SUMMARY:
If tigecycline clearance increases with body size then serum exposure values will be lower in obese class III compared to normal weight subjects because exposure changes inversely with clearance when the dose is fixed without regard to weight.

DETAILED DESCRIPTION:
Not required

ELIGIBILITY:
Inclusion Criteria:

Subjects fulfilling the following criteria will be eligible:

1. males and females, 18 to 50 years of age;
2. non-smoking or light-smoking (≤ 5 cigarettes per day) volunteers;
3. Body mass index: 18.50-24.99 kg/m2 (normal weight) or ≥ 40 kg/m2 (obese class III);
4. female subjects of childbearing potential (self-reported) either surgically sterilized, using an effective method of contraception (diaphragm, cervical cap, condom) or agree to abstain from sex from time of prestudy screening, during entire study period and 1 month following the study period

Exclusion Criteria:

1. history of significant hypersensitivity reaction to any components of Tygacil®;
2. history of significant clinical illness requiring pharmacological management;
3. history of blood donation in the past eight week period;
4. abnormal serum electrolyte or complete blood count requiring further clinical work-up;
5. transaminases (AST or ALT) > 2.5 x upper limit of normal;
6. subjects with stage 4 or 5 chronic kidney disease;
7. positive serum pregnancy test (if female);
8. abnormal electrocardiogram (ECG) as judged by study physician;
9. unable to tolerate venipuncture and multiple blood draws;
10. clinically significant abnormal physical examination defined as a physical finding requiring further clinical work-up;
11. unable to independently provide a written informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manjunath P Pai, PharmD, Principal Investigator — University of Michigan
Locations (1):
- Albany College of Pharmacy, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No
The data have been published as a manuscript J Antimicrob Chemother. 2014 Jan;69(1):190-9.

REFERENCES:
- [Derived] Pai MP. Serum and urine pharmacokinetics of tigecycline in obese class III and normal weight adults. J Antimicrob Chemother. 2014 Jan;69(1):190-9. doi: 10.1093/jac/dkt299. Epub 2013 Jul 23. PMID 23883872

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tigecycline
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tigecycline
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (10.5)
Gender [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Body Mass Index [Median (Full Range); unit: kg/m^2] | 43.8 [20.8 to 53.8]

OUTCOME MEASURES:

1. Primary Outcome: Single-dose Serum AUC of Tigecycline Between Time 0 and 96 Hours
Description: The AUC is the area under the concentration time curve in serum measured in the unit of concentration in milligram of tigeycline per liter of plasma multiplied by the time interval in hours (hour*mg/L)
Time Frame: 4 days (96 hours)
Measure: Mean (Standard Deviation); unit: hour*mg/L
Groups:
- Serum AUC of Tigecycline: All subjects receive a single dose of tigecycline
  Tigecycline: 100 mg IV as a single infusion over 30 minutes
Arm/Group | Serum AUC of Tigecycline
Number analyzed (Participants) | 12
hour*mg/L | 7.64 (1.28)

ADVERSE EVENTS:
Time Frame: 4 days
Arm/Group | Tigecycline
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tigecycline (N=12)
Nausea (Gastrointestinal disorders) | 2 (2)
Emesis (Gastrointestinal disorders) | 1 (1) — Vomitting

LIMITATIONS AND CAVEATS:
Small study sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No